CLINICAL TRIAL: NCT03327987
Title: Safety and Immunogenicity of Influenza Vaccine During the First Post-Transplant Year in Solid Organ Transplant Recipients
Brief Title: Early Flu Shots in SOT
Status: Withdrawn | Type: Observational
Why Stopped: The study was on hold and later withdrawn due to shortage of staff
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 17-5960
Record Dates: First submitted 2017-10-27; First posted 2017-11-01 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Influenza; Solid Organ Transplant
Keywords: vaccine immunogenicity; vaccine safety
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 31-90 days: Patient 31-90 days after transplantation receiving standard of care annual 2017-2018 influenza vaccine.
  Interventions: Biological: standard of care influenza vaccine
- 91-180 days: 91-180 days after transplantation receiving standard of care annual 2017-2018 influenza vaccine.
  Interventions: Biological: standard of care influenza vaccine
- 181-365 days: 181-365 days after transplantation receiving standard of care annual 2017-2018 influenza vaccine.
  Interventions: Biological: standard of care influenza vaccine

INTERVENTIONS:
Biological: standard of care influenza vaccine — The standard of care annual 2017-2018 influenza vaccine will be used for this study.
  Other Names: annual influenza vaccine

SUMMARY:
Although time from transplant has been a factor in vaccine response, there is limited data on immunizations that occur in the first post-transplant year, and there are no data that suggest influenza vaccination early post-transplant may have any adverse effects on the graft. It is suggested that early vaccinations may lead to reduced immunogenicity due to induction immunosuppression. However, not vaccinating patients may leave them vulnerable to influenza infection for a period of time. This study is designed to look at the immunogenicity and side effects of the standard of care influenza vaccine in patients between 31 and 365 days post-transplant.

DETAILED DESCRIPTION:
Influenza virus is an important cause of morbidity in the transplant population and can lead to viral and bacterial pneumonia. Influenza vaccine is effective in the prevention of influenza infection and is recommended by the Canadian National Advisory Committee on Immunization (NACI). The annual influenza vaccine is suggested for transplant patients as the standard of care starting from 3 months post-transplant. Most recent guidelines now suggest that it is reasonable to get a flu shot starting earlier at 1 month post-transplant. Anti-rejection drugs are now tapered more quickly and it is possible that antibodies will be produced against the flu shot as early as 1 month post-transplant. The study hypothesizes that kidney and liver transplant recipients in the early post-transplant period (31-180 days) will have similar immunogenicity as those in the late post-transplant period (>180 days).

ELIGIBILITY:
Inclusion Criteria:

* Kidney, liver or pancreas transplant recipients on at least one immunosuppressive medication
* Age ≥ 18
* Outpatient status
* Greater than 30 days post-transplant

Exclusion Criteria:

* Has already received influenza vaccination for 2017-2018 season
* Egg allergy or allergy to previous influenza vaccine
* Febrile illness in the past one week
* Active Cytomegalovirus viremia
* Use of Rituximab in the past one year
* Ongoing or recent (in past 30 days) therapy for acute rejection
* Chronic kidney insufficiency (creatinine clearance ≤30mL/min or dialysis-dependent
* Previous life-threatening reaction to influenza vaccine (i.e., Guillain Barre Syndrome)
* Receipt of intravenous immunoglobulin (IVIG) in the past 30 days or planning to receive IVIG in the next four weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult solid organ transplant recipients between 31 and 365 days post-transplant.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
Vaccine immunogenicity | 4 weeks
  Vaccine immunogenicity based on assessment of pre- and post-vaccine (4 weeks) antibody titer. A positive vaccine response will be defined based on:
  * Seroconversion rate: serological response with a four-fold or greater increase in HAI antibody titers to each of the three antigens in the vaccine, and
  * Seroprotection rate: HAI titers of ≥1:40 to each of the three antigens post-immunization.

SECONDARY OUTCOMES:
Safety- adverse events | 7 days
  Local and systemic adverse events to vaccination
Safety- graft rejection | 6 months
  Rates of biopsy proven allograft rejection in the 6 months following vaccination
Safety- HLA | 4 weeks
  Development of de novo or increased titer of HLA alloantibody and specifically DSA (donor specific antibody). The 4 weeks post-vaccine sample will be compared with the pre-vaccine samples.
Vaccine efficacy- CMI | 4 weeks
  Analysis of CMI in a subgroup of 60 patients (influenza strain-specific CD4+ and CD8+ T-cell responses; detectable vs. non-detectable and absolute percentage) at four weeks post-vaccine vs. pre-vaccine sample. CMI responses will also be correlated with HAI responses.
Vaccine efficacy- infection | 6 months
  Documented influenza infection (i.e., microbiology proven by the direct fluorescent antibody, viral culture, or PCR) in the six months following vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Deepali Kumar, MD, Principal Investigator — UHN
Locations (1):
- University Health Network, Toronto General Hospital, Multi-Organ Transplant, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No